CLINICAL TRIAL: NCT00130637
Title: Treatment of Active Anterior Uveitis Associated With JIA, Using Humanized Anti-Tac (HAT, Daclizumab)
Brief Title: Human Anti-Tac (Daclizumab) to Treat Juvenile Idiopathic Arthritis (JIA)-Associated Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050208; 05-EI-0208
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Anterior Uveitis; Arthritis, Juvenile Idiopathic; Iritis; Immunosuppression
Keywords: Anterior Uveitis; Arthritis, Juvenile Idiopathic; Daclizumab; Iritis; Immunosuppression; Chronic Inflammatory Eye-Disease; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Uveitis, Anterior; Arthritis, Juvenile; Iritis | interventions — Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daclizumab (Experimental): IV daclizumab
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Daclizumab
  Other Names: Human Anti-Tac

SUMMARY:
This study will examine the safety and effectiveness of a monoclonal antibody called humanized anti-Tac (HAT, also called daclizumab) to treat children and adolescents with uveitis (chronic inflammatory eye disease) associated with juvenile idiopathic arthritis (JIA). Monoclonal antibodies are genetically engineered proteins made in large quantities and directed against a specific target in the body. The HAT antibody is designed to prevent a specific chemical interaction needed for immune cells to produce inflammation. Current treatments for uveitis include steroids and immune-suppressing drugs. These treatments do not always work or they may cause significant side effects. This study will determine whether daclizumab can improve uveitis in children and reduce the need for other medicines.

Patients between 6 and 18 years of age with active non-infectious JIA-associated uveitis requiring treatment with anti-inflammatory medications as often as three times a day or more may be eligible for this study.

Each candidate is screened with a medical history, physical examination, blood tests, eye examination, and the following specialized tests:

* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating the presence of inflammation.
* Optical coherence tomography to measure retinal thickness. The eyes are examined through a machine that produces cross-sectional pictures of the retina. These measures are repeated during the study to determine changes, if any, in retinal thickening.
* Stereoscopic color fundus photography to examine the back of the eye. The pupils are dilated with eye drops to examine and photograph the back of the eye.

Upon entering the study, participants receive a 90-minute infusion of daclizumab through a catheter (plastic tube) placed in an arm vein. They return to the clinic after 14 days and again after 28 days for repeat eye examinations, blood tests, and daclizumab infusions. Four weeks after the third infusion, patients are examined for response to treatment. Those who have benefited from daclizumab may continue receiving monthly infusions of the drug for up to one year. A blood test and eye examination are done at the time of each infusion. Patients whose disease has remained active 12 weeks after the first infusion are taken off the study and treated with other medications.

DETAILED DESCRIPTION:
Pediatric uveitis represents 5-10 % of all patients with uveitis. Uveitis refers to intraocular inflammatory diseases. The most common type of non-infectious pediatric uveitis, associated with a systemic disease, is JIA-associated chronic, anterior uveitis. Therapeutic considerations for pediatric uveitis are often very challenging. Current therapeutic modalities include corticosteroids and other immunosuppressive agents. These modalities are not always effective at controlling the disease. In addition they can also be associated with a higher rate of ocular side effects. To further add to this challenge, pediatric uveitis has a higher rate of ocular complications, even with the current therapies. Consequently, an effective treatment with a safer side effect profile is highly desirable. Daclizumab is a humanized monoclonal antibody directed against the high affinity interleukin-2 (IL-2) receptor CD25 or Tac subunit. The IL-2 receptor system plays a central role in mediating immune responses. Blocking this system impedes immune responses and can inhibit local inflammatory responses, including uveitis. Pilot studies using intravenous or subcutaneous daclizumab treatments suggest that daclizumab treatments at 2 mg/kg every 2-4 weeks for quiescent uveitis may effectively replace the other immunosuppressive medications in a majority of cases.

Because we have little experience using daclizumab for active uveitis in a pediatric population, this feasibility study will enroll seven study participants that would normally be treated with systemic, high-dose corticosteroids or other cytotoxic, systemic immunosuppressive medications. Since daclizumab for other indications can be tolerated with repeated dosing at 8-10 mg/kg, we will administer daclizumab to reach high serum levels with a pair of doses at 8 mg/kg and 4 mg/kg two weeks apart. The primary objective of this study is to collect preliminary information on the utility of acute daclizumab therapy on active ocular inflammation in a pediatric population. The primary outcome is resolution of active disease defined as a two step reduction in the anterior chamber cell scale from baseline. Safety assessment will be made at 28 days and efficacy assessment at 8 weeks after the initial daclizumab injection. Secondary outcomes will include fluorescein retinal vascular leakage, cystoid macular edema, vitreous haze and visual acuity. In addition all adverse events will be collected regardless of possible relation to daclizumab. Participants who do not meet the safety end point at day 28 will be permitted to continue IV daclizumab maintenance treatments beginning at Day 28 with 2 mg/kg every 4 weeks. An efficacy assessment will be made at 8 weeks, and patients who show a 2 step reduction in their intraocular inflammation, and has not met the safety end point, will continue daclizumab treatment with 2mg/kg every 4 weeks for a total of 52 weeks in the study. At any time during the follow-up period, if a participant loses greater than 3 lines of visual acuity from baseline study, or meet the safety end point, treatments will be discontinued.

The primary objective of this feasibility study is to gain preliminary information regarding the safety and possible efficacy of daclizumab to treat active uveitis, associated with JIA.

The primary focus of this feasibility study is a short or acute response trial to relatively high-dose daclizumab infusions to observe if the anterior cell and flare associate with active JIA-associated uveitis can be promptly reduced. In order to qualify for enrollment, each participant must meet all of the inclusion criteria and not meet any of the exclusion criteria. This study will enroll seven participants at the National Eye Institute (NEI) who currently have active JIA-associated active uveitis. Enrollment is expected to take approximately three months. The two induction treatments will be completed within 14 days, with the primary safety evaluation at Day 14 and Day 28 and primary efficacy assessment at 12 weeks. An induction regimen of intravenous (IV) daclizumab at 8 mg/kg is given on Day 0 followed by another IV dose of 4 mg/kg at Day 14, provided the safety endpoint has not been met.

An efficacy assessment will be made at 12 weeks, and patients who show a 2-step reduction in their intraocular inflammation, and has not met the safety endpoint, will continue with daclizumab therapy. Meeting the safety failure criterion or having a serious adverse affect attributable to the daclizumab therapy will be cause for termination from further daclizumab study treatments. Continuing follow-up and standard-of-care alternative treatments with a potentially reduced visit schedule will be provided through the duration of the trial if daclizumab treatments are suspended. After the trial, participants may seek other standard-of-care treatments from their own physician or ophthalmologist or they may be eligible to enroll in other research trials if these are available.

Participants who show a 2-step reduction in their ocular inflammation or a decrease to inactivity, without serious adverse events, will have the option to receive extended treatments of 2 mg/kg IV daclizumab treatments at 4-week intervals, beginning day 28, for up to a total of 52 weeks in the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant is from 6 to 18 years of age, inclusive;
  2. Participant has a diagnosis of non-infectious uveitis associated juvenile idiopathic arthritis (JIA) requiring treatment to control their intraocular inflammatory disease with anti-inflammatory medications, systemic and/or topical at high frequency intervals (greater than or equal to 3 times a day).
  3. Participant's uveitis is considered active on current regimen
  4. Participant has uveitis with at least a grade of 1+ for anterior chamber cells in at least one eye
  5. Participant's uveitis is currently treated or untreated at the time of enrollment
  6. Participant has visual acuity in at least one eye of 20/640 or better (Early Treatment Diabetic Retinopathy Study (ETDRS) or Electronic Visual Acuity-Amblyopia Treatment Study (EVA-ATS), log minimum angle of resolution (logMAR) less than 1.54).
  7. Participant has normal renal or liver function or evidence of no worse than mild abnormalities as defined by the "Common Toxicity Criteria for Adverse Events" (CTCAE) version 3.0, including:

     Test Parameter Age (yrs) Pediatric Mild Limit

     Serum creatinine 6-12 1.0 mg/dL

     13-18 1.6 mg/dL

     Proteinuria 6-18 3 g/L

     Uric acid 6-18 9.9 mg/dL

     Blood Urea Nitrogen (BUN) 6-18 2.0 upper normal limit

     Aspartate aminotransferase (Serum glutamic-oxaloacetic transaminase) (AST (SGOT)) 6-18 2.5 upper normal limit

     Alanine aminotransferase (Serum glutamic pyruvic transaminase) (ALT (SGPT)) 6-18 2.5 upper normal limit
  8. Participant agrees not to undergo elective ocular surgery (e.g., cataract extraction) for the first 6 months of the study.
  9. Participant has an absolute neutrophil count above 750.
  10. Participant is not currently pregnant or lactating.
  11. Participant with reproductive potential and who is sexually active agrees to use acceptable birth control methods throughout the course of the study and for 6 months after completion of treatment.
  12. All participants at enrollment has a parent or legal guardian who is able to understand and sign a consent form on their behalf before entering into the study, and participant signs an assent as a minor.
  13. Meet American College of Rheumatology Criteria for Juvenile Rheumatoid Arthritis (JRA)/JIA (Appendix) but is not newly diagnosed, and has had systemic treatment for their uveitis.
  14. Be able to undergo slit lamp biomicroscopy for assessment of anterior chamber cells.
  15. Be able to comply with the study requirements.
  16. Be up to date on all recommended childhood immunizations.

EXCLUSION CRITERIA:

1. Participants under the age of 6 years will not be enrolled in the study due to the reported higher incidence of adverse events related or unrelated to the administration of daclizumab in post-transplant pediatric studies compared to children over age 6.
2. Participants who had received previous treatment with an IL-2 directed monoclonal antibody or any other investigational agent that would interfere with the ability to evaluate the safety, efficacy or pharmacokinetics of daclizumab.
3. Participants with a history or diagnosis of Behcet's disease.
4. Participant has a significant active infection.
5. Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past 5 years.
6. Participant has used latanoprost (Xalatan) within two weeks prior to study enrollment or has a likely need.
7. Participant for whom administration of fluorescein dye is medically contraindicated.
8. Have a media opacity that precludes assessment of anterior chamber inflammation.
9. Be a female who is pregnant or lactating.
10. Refuse to use contraception during the study and 6 months after termination of active study therapy, if child-bearing or fathering potential exists.
11. Have active serious infections or a history of recurring serious infections.
12. Evidence of spondyloarthropathy or enthesopathy.
13. Have active joint or systemic inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chylack LT Jr. The ocular manifestations of juvenile rheumatoid arthritis. Arthritis Rheum. 1977 Mar;20(2 Suppl):217-23. PMID 263899
- [Result] Sen HN, Levy-Clarke G, Faia LJ, Li Z, Yeh S, Barron KS, Ryan JG, Hammel K, Nussenblatt RB. High-dose daclizumab for the treatment of juvenile idiopathic arthritis-associated active anterior uveitis. Am J Ophthalmol. 2009 Nov;148(5):696-703.e1. doi: 10.1016/j.ajo.2009.06.003. Epub 2009 Aug 6. PMID 19664754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: single center, 6 participants
Pre-assignment Details: pilot, non-randomized, open-label trial
Groups:
- Daclizumab: An induction regimen of intravenous (IV) daclizumab at 8 mg/kg was given on Day 0 followed by another IV dose of 4 mg/kg at Day 14, provided the safety endpoint was not met. Participants who showed a two-step reduction in their ocular inflammation or a decrease to inactivity, without serious adverse events, had the option to receive extended treatments of 2 mg/kg IV daclizumab treatments at 4-week intervals, beginning day 28, for up to a total of 52 weeks.
Period: Overall Study
Arm/Group | Daclizumab
Started | 6
Completed | 3
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daclizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Two-step Reduction in Inflammation
Description: Number of participants with a two-step reduction (or down to 0 out of a scale of 0 to 4+) of anterior chamber (AC) inflammation according to Standardization of Uveitis Nomenclature (SUN) criteria, while on a topical corticosteroid schedule of less than 3 times a day. Grade 0 is the best score on this scale with <1 cell in the field and 4+ is the worst score on this scale with >50 cells in the field.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Daclizumab
Number analyzed (Participants) | 6
participants | 5

2. Primary Outcome: Number of Participants Reporting a Serious Adverse Event (SAE)
Description: Safety of acute daclizumab use in JIA-associated uveitis was assessed through serious adverse events (SAE).
Time Frame: 52 weeks
Measure: Number; unit: participant
Arm/Group | Daclizumab
Number analyzed (Participants) | 6
participant | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 52 week study period
Description: Event descriptions were not mapped to a standardized term. General disorders was chosen as the organ system for events categorized as "Other" or "Pain".
Arm/Group | Daclizumab
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daclizumab (N=6)
palpitations (Cardiac disorders) | 1 (1) — palpitations with normal echocardiogram (ECG), patient hospitalized for observation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daclizumab (N=6)
herpes zoster skin infection (Infections and infestations) | 1 (1) — Verbatim event description reported by site staff was "maculopapular rash (positive for varicella virus)"
lower extremity edema (General disorders) | 1 (1) — Verbatim event description reported by site staff was "bilateral ankle swelling and associating pain". This event was secondary to naproxen as it resolved upon discontinuation of naproxen
Allergy symptoms (Immune system disorders) | 1 (1)
Ankle stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Aphtous ulcer on right lower gum (General disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Bilateral Hand and wrists inflammation, Mild Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cold Symptoms/Sore throat (Infections and infestations) | 1 (1)
Decreased appetite with associated nausea (Gastrointestinal disorders) | 1 (1)
Decreased Hgb and Hct (Blood and lymphatic system disorders) | 1 (1)
Elevated AST (Metabolism and nutrition disorders) | 3 (3)
Elevated Cholesterol level (Metabolism and nutrition disorders) | 1 (1)
Elevated CPK (Metabolism and nutrition disorders) | 1 (1)
Elevated ESR (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated potassium level (Metabolism and nutrition disorders) | 1 (1)
Elevated Urine WBC (Renal and urinary disorders) | 1 (1)
Elevated WBC (Blood and lymphatic system disorders) | 2 (2)
Erythematous area of Lower Eyelid (General disorders) | 1 (1)
Stomach virus (Infections and infestations) | 1 (1)
Gum abscess (Infections and infestations) | 1 (1)
Headache (General disorders) | 1 (1)
Headaches/Back Pain (General disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (1)
Knee Pain (General disorders) | 1 (1)
Low Hgb and Hct (Blood and lymphatic system disorders) | 2 (2)
Low platelets (Blood and lymphatic system disorders) | 1 (1)
Low White Blood Count (Blood and lymphatic system disorders) | 1 (1)
Mild myalgia in legs (General disorders) | 1 (1)
Mild pain left knee and hip after playing soccer. (General disorders) | 1 (1)
mild right shoulder pain (General disorders) | 1 (1)
Mild shoulder pain (General disorders) | 1 (1)
Mouth Sores (General disorders) | 1 (2)
Mucous membrane Ulcers (General disorders) | 1 (1)
Nasal congestion causing right ear pain (Infections and infestations) | 1 (1)
Neck and Lower back pain (General disorders) | 1 (1)
Nose bleed (Blood and lymphatic system disorders) | 1 (1)
Occasional dysuria (Renal and urinary disorders) | 1 (1)
Occasional Light headiness (Cardiac disorders) | 1 (1)
Pain Right great toe (General disorders) | 1 (1)
Painful Right Wrist (General disorders) | 1 (1)
Persistent cough (Infections and infestations) | 1 (1)
Photophobia (General disorders) | 1 (1)
Planter tenderness (Hepatobiliary disorders) | 1 (1)
Pustules over abdominal area (Infections and infestations) | 1 (1)
Right knee pain without inflammation (General disorders) | 1 (1)
Right Thumb sore and swollen (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Knee Pain few hrs after prolonged exertion (General disorders) | 1 (1)
Runny Nose (Infections and infestations) | 1 (1)
Ruptured blister inner lower lip (Gastrointestinal disorders) | 1 (1)
Rash (Infections and infestations) | 1 (1) — Verbatim event description reported by site staff was "scabies, rash chest, under arms and inner thighs"
Slight increase in total bilirubin (Metabolism and nutrition disorders) | 1 (1)
Slightly Swollen right anterior pilla of tonsil (General disorders) | 1 (1)
Sore Throat, fever, body ache (Infections and infestations) | 1 (1)
Sore Throat, Low grade fever, Malaise (Infections and infestations) | 1 (1)
Squinting OU (Eye disorders) | 1 (1)
Stomach Flu (Infections and infestations) | 1 (1)
Stuffy Nose and Sore Throat (Infections and infestations) | 1 (1)
Systemic Joint Inflammation, & assoc. joint pain. (Musculoskeletal and connective tissue disorders) | 1 (1)
Tonsilitis with associated fever (Infections and infestations) | 1 (1)
Tooth Extraction (General disorders) | 1 (1)
Slight Leukocyte esterase increase (Renal and urinary disorders) | 1 (1)
Upper respiratory Infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Throat infection (Infections and infestations) | 1 (1)
Slight cold (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
The results of this trial need to be interpreted cautiously because of the small number of patients, the heterogeneity of the patient population (such as one participant with systemic JIA), and the nonrandomized and unmasked nature of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No